CLINICAL TRIAL: NCT04338828
Title: Nitric Oxide Inhalation Therapy for COVID-19 Infections in the Emergency Department
Brief Title: Nitric Oxide Inhalation Therapy for COVID-19 Infections in the ED
Acronym: NO COV-ED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Absence of patients meeting criteria following initial COVID surge. DMSB recommended analysis of results to date and early closure.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, N. Stuart Harris MD MFA, Principal Investigator, Division Chief of Wilderness Medicine, Department of Emergency Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P00XXXX
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: COVID19
Keywords: inhaled nitric oxide; emergency department; emergency medicine; respiratory infection
MeSH Terms: conditions — COVID-19; Emergencies; Respiratory Tract Infections | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Inhaled nitric oxide
  Interventions: Drug: Nitric Oxide Gas
- Control Group (Placebo Comparator): Inhaled supplemental oxygen
  Interventions: Other: Inhaled Supplemental Oxygen

INTERVENTIONS:
Drug: Nitric Oxide Gas — Inhaled NO administered at target inspired concentration 140 - 300 ppm for 20-30 minutes
  Arms: Treatment Group
Other: Inhaled Supplemental Oxygen — 2 L/min oxygen therapy
  Arms: Control Group

SUMMARY:
The spread of novel Coronavirus (2019-nCoV) related infection (COVID-19) has led to many patient presentations in the emergency department for respiratory complaints, with many of these patients requiring ICU admission and ventilatory support. While COVID-19 patients have an increased need for supportive care, there is currently no specific treatment directed against 2019-nCoV. Nitric oxide inhalation has been used as a pulmonary vasodilator and has been found to have antiviral activity against other coronavirus strains. The primary aim of this study is to determine whether inhaled NO improves short term respiratory status, prevents future hospitalization, and improves the clinical course in patients diagnosed with COVID-19 specifically in the emergency department.

DETAILED DESCRIPTION:
The spread of novel Coronavirus (2019-nCoV) related infection (COVID-19) has led to many patient presentations in the emergency department for respiratory complaints, with many of these patients requiring ICU admission and ventilatory support. While COVID-19 patients have an increased need for supportive care, there is currently no specific treatment directed against 2019-nCoV. Nitric oxide inhalation has been used as a pulmonary vasodilator and has been found to have antiviral activity against other coronavirus strains.

Preliminary data support a microbicidal effect of high concentration inhaled NO. We hypothesize that high concentration inhaled NO can have a viricidal effect against SARS-Cov-2 and prevent the deterioration to a severe form of COVID-19 when administered at an early stage of the disease. Additional potential mechanisms why INO may be effective in this indication: 1)improves V/Q ratio, 2) reduces PVR and PAP, 3) Anti-thrombotic in lung. This would have potential benefit for the patients in terms of reducing the severity of the clinical course and time to recovery. An additional benefit could be for the society since a faster and a less severe clinical course could protect limited hospital resources (ED, floor, and ICU) from being overwhelmed.

The primary aim is to prevent the deterioration of mild COVID-19 infection (defined by a RT-PCR positive for SARS-CoV-2 in a specimen from any site) with respiratory signs/ symptoms to a more severe form of the disease as defined by the patient needing to 1) return to the ED, 2) be admitting to the hospital, 3) be intubated, 4) and all cause 28 day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Presentation to the ED with respiratory symptoms likely caused by COVID-19
* Patient displays at least one of the following

  1. respiratory rate ≥ 24
  2. new cough
  3. new atypical chest pain
  4. new dyspnea
  5. oxygen saturation < 97% at rest
  6. chest x-ray with new changes consistent with COVID-related airspace disease
* Cleared for discharge home by attending physician
* Obtained COVID testing (results not required at time of enrollment)
* Onset of symptoms ≤12 days prior to ED visit

Exclusion Criteria:

* Attending physician estimation (< 50% likelihood) of other more likely non-COVID etiology
* Presence of tracheostomy
* Requirement of oxygen therapy to maintain resting oxygen saturation of > 94%
* Clinical contraindication to use of inhaled nitric oxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Rates of return visits to the ED | 28 days
  Difference within treatment and control groups with COVID-related symptoms/disease in their likelihood to return to the ED with worsening symptoms

SECONDARY OUTCOMES:
Inpatient hospitalizations required | 28 days
  Difference within treatment and control groups with COVID-related symptoms/disease in their likelihood to require hospitalization during their COVID-19 course
Rates of intubation | 28 days
  Difference within treatment and control groups with COVID-related symptoms/disease in their likelihood to require intubation during their COVID-19 course
Rates of mortality | 28 days
  Difference within treatment and control groups with COVID-related symptoms/disease in their likelihood to die of any cause within 28 days of their initial ED visit

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No